CLINICAL TRIAL: NCT00749606
Title: Weight Loss in Primary Care: a Translation of the Diabetes Prevention Program
Brief Title: Study to Promote Weight Loss in Primary Care Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ruth Weinstock, Principal Investigator, State University of New York - Upstate Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R18DK078553 (NIH); R18DK078553 (NIH)
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Results first posted 2017-12-05 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Obesity
Keywords: Obesity; Metabolic syndrome; Weight loss; Diabetes prevention
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual Telephone Intervention (Experimental): Individually administered weight loss intervention, based on the Diabetes Prevention Program, delivered by telephone in primary care practices.
  Interventions: Behavioral: Individual telephone intervention
- Group Telephone Intervention (Active Comparator): Group education conference calls to deliver the weight loss intervention, based upon the Diabetes Prevention Program, in primary care practices.
  Interventions: Behavioral: Group telephone intervention

INTERVENTIONS:
Behavioral: Individual telephone intervention — Individually administered telephone-based weight loss intervention based on the Diabetes Prevention Program (weekly nurse calls for the first 5 weeks, then monthly, to cover the 16 topics from the Diabetes Prevention Program). In year 1 (after the first 5 weeks), the "coach" will have 3 weekly calls per month with participants. Contact will decrease to monthly in year 2. In year 3 there will be no contact arranged by study staff.
  Arms: Individual Telephone Intervention
Behavioral: Group telephone intervention — Group education conference calls administered weight loss intervention based on the Diabetes Prevention Program (weekly nurse calls for the first 5 weeks, then monthly, to cover the 16 topics from the Diabetes Prevention Program). In year 1 (after the first 5 weeks), the "coach" will have 3 weekly calls per month with participants. Contact will decrease to monthly in year 2. In year 3 there will be no contact arranged by study staff.
  Arms: Group Telephone Intervention

SUMMARY:
The purpose of this study is to determine if primary care based, telephone-delivered weight loss interventions are effective.

DETAILED DESCRIPTION:
Obesity is related to the rising incidence of type 2 diabetes. Cost-effective interventions leading to sustained weight loss are needed to improve the public health and reverse the alarming rise in diabetes, its cardiovascular complications and other obesity-related illnesses. The Diabetes Prevention Program is identified as a model for a successful weight loss intervention. The proposed study is a randomized controlled trial of 2 active telephone-based interventions based on the Diabetes Prevention Model that will be delivered at primary care sites.

ELIGIBILITY:
Inclusion Criteria:

* Obese
* Metabolic syndrome
* Read and write English
* Planning to stay in treatment with their PCP for the next 3 years
* On stable doses of medications for chronic diseases such as hypothyroidism for 3 years

Exclusion Criteria:

* Unstable health
* Diabetes mellitus
* Severe medical comorbidities that might interfere with their ability to participate in intervention such as severe psychiatric disease or significant heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2009-06; Primary Completion 2012-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth S. Weinstock, MD PhD, Principal Investigator — State University of New York - Upstate Medical University; Paula Trief, PhD, Principal Investigator — State University of New York - Upstate Medical University

REFERENCES:
- [Result] Weinstock RS, Trief PM, Cibula D, Morin PC, Delahanty LM. Weight loss success in metabolic syndrome by telephone interventions: results from the SHINE Study. J Gen Intern Med. 2013 Dec;28(12):1620-8. doi: 10.1007/s11606-013-2529-7. Epub 2013 Jul 11. PMID 23843020
- [Result] Trief PM, Cibula D, Delahanty LM, Weinstock RS. Depression, stress, and weight loss in individuals with metabolic syndrome in SHINE, a DPP translation study. Obesity (Silver Spring). 2014 Dec;22(12):2532-8. doi: 10.1002/oby.20916. Epub 2014 Sep 24. PMID 25251749
- [Result] Trief PM, Weinstock RS, Cibula D, Delahanty LM. Sustained weight loss one year after group telephone intervention: 3-year results from the SHINE study. Diabetes Res Clin Pract. 2014 Dec;106(3):e74-8. doi: 10.1016/j.diabres.2014.09.032. Epub 2014 Oct 5. PMID 25451907
- See also: Weight Loss Success in Metabolic Syndrome by Telephone Interventions: Results from the SHINE Study. — http://www.ncbi.nlm.nih.gov/pubmed/23843020

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment took place from June 22, 2009 - Oct 2, 2010 from 5 diverse primary care practice sites in upstate NY: Oneida Healthcare Center (small city), Pulaski Health Center (rural), Syracuse Community Healthcare Center and University Health Care Center (urban, poor, medium city), and University Internists (higher income, medium city).
Groups:
- Individual Calls: Individually administered weight loss intervention, based on the Diabetes Prevention Program, delivered by telephone in primary care practices.
  Individual telephone intervention: Individually administered telephone-based weight loss intervention based on the Diabetes Prevention Program (weekly nurse calls for the first 5 weeks, then monthly, to cover the 16 topics from the Diabetes Prevention Program). In year 1 (after the first 5 weeks), the "coach" will have 3 weekly calls per month with participants. Contact will decrease to monthly in year 2. In year 3 there will be no contact arranged by study staff.
- Conference Calls: Group education conference calls to deliver the weight loss intervention, based upon the Diabetes Prevention Program, in primary care practices.
  Group telephone intervention: Group education conference calls administered weight loss intervention based on the Diabetes Prevention Program (weekly nurse calls for the first 5 weeks, then monthly, to cover the 16 topics from the Diabetes Prevention Program). In year 1 (after the first 5 weeks), the "coach" will have 3 weekly calls per month with participants. Contact will decrease to monthly in year 2. In year 3 there will be no contact arranged by study staff.
Period: Year 1
Arm/Group | Individual Calls | Conference Calls
Started | 129 | 128
Completed | 74 | 80
Not Completed | 55 | 48
Period: Year 2
Arm/Group | Individual Calls | Conference Calls
Started | 74 | 80
Completed | 63 | 72
Not Completed | 11 | 8
Period: Year 3 (Observation)
Arm/Group | Individual Calls | Conference Calls
Started | 63 | 72
Completed | 63 | 69
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individual Calls | Conference Calls | Total
Number analyzed (Participants) | 129 | 128 | 257
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (13.1) | 52.7 (12.8) | 51.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 65 | 166
  Male | 28 | 63 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 128 | 126 | 254
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 15 | 33
  White | 110 | 112 | 222
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 129 | 128 | 257
Weight [Mean (Standard Deviation); unit: kg] | 105.8 (23.6) | 109.4 (26.1) | 107.6 (24.9)

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: Weight (kg)
Time Frame: baseline, 1, 2, 3 years
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Individual Calls | Conference Calls
Number analyzed (Participants) | 129 | 128
kg
  Baseline | 105.8 (23.6) | 109.4 (26.1)
  Year 1 | 102.07 (19.73) | 101.23 (18.97)
  Year 2 | 104.20 (21.57) | 100.33 (20.49)
  Year 3 | 104.47 (21.51) | 100.27 (20.44)
Statistical Analysis 1: Comparison: Individual Calls vs Conference Calls; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; Mixed linear models analyzed within-subject variation in repeated measures over time. Intention to treat analysis used 5 imputations for missing data

2. Secondary Outcome: Blood Pressure
Description: Systolic blood pressure (mm Hg) / Diastolic blood pressure (mm Hg)
Time Frame: baseline, 1, 2, 3 years
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Individual Calls | Conference Calls
Number analyzed (Participants) | 129 | 128
mmHg
  Systolic blood pressure baseline | 128.75 (31.13) | 129.54 (31.24)
  Systolic blood pressure Year 1 | 129.94 (41.83) | 129.90 (40.48)
  Systolic blood pressure Year 2 | 132.05 (45.59) | 132.60 (43.50)
  Systolic blood pressure Year 3 | 134.43 (45.06) | 131.17 (43.04)
  Diastolic blood pressure Baseline | 75.24 (15.93) | 75.61 (16.00)
  Diastolic blood pressure Year 1 | 76.23 (21.33) | 74.83 (20.63)
  Diastolic blood pressure Year 2 | 77.85 (23.24) | 76.73 (22.18)
  Diastolic blood pressure Year 3 | 78.16 (23.00) | 75.74 (21.95)

3. Secondary Outcome: Fasting Lipid Panel
Description: LDL-cholesterol (mg/dL)
Time Frame: baseline, 1, 2, 3 years
Population: Note: LDL-cholesterol measurements were not available for 13 participants in the Individual Call arm and 6 participants in the Conference Call arm
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Individual Calls | Conference Calls
Number analyzed (Participants) | 116 | 122
mg/dL
  Baseline | 107.32 (51.17) | 108.01 (49.91)
  Year 1 | 113.21 (68.81) | 109.11 (66.94)
  Year 2 | 113.80 (75.97) | 107.91 (72.13)
  Year 3 | 109.74 (75.21) | 107.02 (72.10)

4. Secondary Outcome: Fasting Glucose Level
Description: Fasting glucose (mg/dL)
Time Frame: baseline, 1, 2, 3 years
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Individual Calls | Conference Calls
Number analyzed (Participants) | 129 | 128
mg/dL
  Baseline | 99.70 (30.05) | 99.44 (30.19)
  Year 1 | 100.43 (40.21) | 100.72 (39.15)
  Year 2 | 101.12 (43.83) | 101.37 (41.84)
  Year 3 | 101.39 (43.42) | 100.61 (41.46)

5. Secondary Outcome: Health Behaviors (Diet, Physical Activity)
Description: National Cancer Institute Fat screener
Time Frame: baseline, 6 months, 1 and 2 years
Measure: Mean (Standard Error); unit: percentage of daily calories from fat
Arm/Group | Individual Calls | Conference Calls
Number analyzed (Participants) | 129 | 128
percentage of daily calories from fat
  Change from baseline at 6 months | 2.644 (0.622) | 1.392 (0.617)
  Change from baseline at 1 year | 2.910 (0.599) | 1.402 (0.605)
  Change from baseline at 2 years | 1.173 (0.643) | 1.395 (0.632)

6. Secondary Outcome: SF-12 Physical Summary Score
Description: The impact of physical health on overall quality of life; higher score reflects better quality of life. Range 0-100 (0 indicates the lowest level and 100 the highest level of health).
Time Frame: baseline, 6 months, 1 and 2 years
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Individual Telephone Intervention | Group Telephone Intervention
Number analyzed (Participants) | 129 | 128
units on a scale
  Change from baseline at 6 months | 2.543 (1.056) | 1.274 (1.028)
  Change from baseline at 1 year | 1.064 (1.200) | 1.082 (1.102)
  Change from baseline at 2 years | 1.506 (1.358) | 0.932 (1.297)

7. Secondary Outcome: International Physical Activity Questionnaire
Description: Measure of physical activity is calculated as in mets/week
Time Frame: baseline, 6 months, 1 and 2 years
Measure: Mean (Standard Error); unit: mets per week
Arm/Group | Individual Calls | Conference Calls
Number analyzed (Participants) | 129 | 128
mets per week
  Change from baseline at 6 months | -0.611 (3.781) | 8.427 (3.717)
  Change from baseline at 1 year | 7.229 (3.978) | 11.812 (3.735)
  Change from baseline at 2 years | 10.099 (4.976) | 15.968 (4.646)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Individual Calls | Conference Calls
Serious Adverse Events (participants affected / at risk) | 19/129 | 16/128
Other Adverse Events (participants affected / at risk) | 0/129 | 0/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individual Calls (N=129) | Conference Calls (N=128)
Hospitalization (Cardiac disorders) | 2 (2) | 4 (5)
Hospitalization (Psychiatric disorders) | 1 (1) | 1 (2)
Hospitalization (Endocrine disorders) | 1 (1) | 0 (0)
Hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hospitalization (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hospitalization (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hospitalization (General disorders) | 3 (3) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Hospitalization (Vascular disorders) | 1 (1) | 2 (2)
Hospitalization (Immune system disorders) | 0 (0) | 1 (1)
Hospitalization (Infections and infestations) | 2 (2) | 4 (4)
Hospitalizations (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hospitalization (Surgical and medical procedures) | 7 (7) | 5 (6)
Hospitalization (Nervous system disorders) | 3 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No